CLINICAL TRIAL: NCT07134634
Title: Effekt Eines Vibrierenden Therapieballs Auf Den Tremor Und Alltagsaktivitäten Bei PatientInnen Mit Verschiedenen Tremorsyndromen
Brief Title: Effect of a Vibrating Therapy Ball on Tremor and Daily Activities in Patients With Different Tremor Syndroms
Status: Recruiting | Type: Observational
Sponsor: Parkinson's Clinic in Beelitz-Heilstatten (Other)
Responsible Party: Principal Investigator, PD Dr. med.habil. Doreen Gruber, Principal Investigator, Parkinson's Clinic in Beelitz-Heilstatten
Other Study IDs: 2024-103-BO-ff
Record Dates: First submitted 2025-03-05; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
Keywords: Tremor
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- tremor cohort
  Interventions: Device: tremor device

INTERVENTIONS:
Device: tremor device — tremor ball on versus tremor ball off

SUMMARY:
Tremors, e.g. in patients with Parkinson's disease and essential tremor, are often pharmacoresistant, meaning that invasive treatment options such as deep brain stimulation are used at an early stage. Sufficient complementary non-pharmacological treatment alternatives do not yet exist. Patients with tremor are often severely restricted in their ability to carry out everyday activities and require support from relatives and carers, e.g. with food intake and hygiene measures.

The VILIM ball device is a CE-certified, non-invasive, portable physiotherapeutic aid. It is intended for use at home or in a professional setting as a mechanical vibration therapy device to temporarily reduce hand tremor.

With this vibrating therapy ball (VILIM tremor ball), which is customised to the patient's tremor during a training phase, should temporarily reduce tremor by up to 50%, according to the manufacturer. The effect can last up to 4 hours, so that patients should be able to carry out their everyday activities better, e.g. eating, writing, etc. (https://vilimed.com).

An initial study already reported a reduction in tremor in patients with Parkinson's disease and essential tremor. However, this study lacked a training phase, a control group and an examination of the effect on functions relevant to everyday life, meaning that reliable conclusions on the effect are only possible to a limited extent In this study, the influence of the portable physiotherapeutic therapy device (VILIM ball) on tremor in the upper extremity compared to an alternative therapy as a control condition in patients with Parkinson's tremor, essential tremor and other tremor syndromes will be investigated for the first time. The evaluation of the physician-associated scales will additionally be carried out by an independent physician in a single-blinded manner on the basis of video documentation.

The primary endpoint is a significant effect of the therapy ball on tremor, quantified and qualified using Clinical Global Impression Severity (CGI severity:

Assessment by doctor and patient) and validated disease-specific tremor scales: MDS-UPDRS IIl including the Tremor subscale, TETRAS between tremor ball therapy (Ball-On) alternative therapy (Ball-Off). Secondary endpoints include the effect of the therapy ball compared to the ball-off condition on tremor analysis data (e.g. frequency peak, amplitude) of an accelerometer, mini darts, writing tasks, specific tasks of daily life: e.g. bringing a spoon with liquid to the mouth, pouring water into a glass without losing the liquid and the success of the therapy using CGI improvement (doctor and patient).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of tremor
2. ability to complete the tests
3. no cognitive deficits relevant to everyday life

Exclusion Criteria:

1. cognitive deficits relevant to everyday life that influence therapy
2. pronounced dystonia, dyskinesia
3. Pregnancy
4. Acute thrombotic process (myocardial infarction, (acute vascular constriction)
5. Implants in activated regions of the body (e.g.artificial joints)
6. Acute inflammation of the locomotor system active arthrosis or arthropathy e.g. acute inflammationor swelling of joints

   * Acute tendinopathy in activated regions of the body (acute tendon inflammation)

     • Acute desmopathy (acute problems at the intervertebral disc)
   * Fresh fractures in activated regions of the body
7. Post-surgery wounds and fresh wounds in activated regions of the body or incomplete wound healing
8. Rheumatoid arthritis
9. Epilepsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with different tremor syndroms
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The effect of the vibrating therapy ball on hand tremor will be assessed before and after use, comparing ball-on vs. ball-off. The following scores will be used: | 2 years
  Primary endpoints:
  * Change in Clinical Global Impression Severity (Assessment by physician and patient) after using the therapy ball (Score 0 to 7 pts., a lower score means better outcome)
  * Change in MDS-UPDRS part IIl (Score 0 - 132 pts., a lower score means a better outcome)
  * Change in 2 items of TETRAS Activities of Daily Living Subscale (Score 0 -8 pts., a lower score means a better outcome)
  Secondary endpoints:
  * Changes in the frequency of the tremor (in Hz) using an acceleromter. A lower value means a better outcome
  * Changes in amplitude of the tremor (in mm) using an accelerometer. A lower value means a better outcome
  * changes in 3 items of Fahn-Tolosa-Marin-Tremor-Rating-Scale (0-12 pts.). A lower score means a better outcome
  * Change in Clinical Global Impression-Improvment Scale (CGI-I), (0-7 pts., lower score means better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- ParkinsonBeelitzHeilstaetten, Beelitz, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Following the data publication, IPD will be available from the coresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: see above
Access Criteria: see above

REFERENCES:
- [Background] Haubenberger D, Hallett M. Essential Tremor. N Engl J Med. 2018 May 10;378(19):1802-1810. doi: 10.1056/NEJMcp1707928. No abstract available. PMID 29742376
- [Background] Abramavicius S, Venslauskas M, Vaitkus A, Gudziunas V, Laucius O, Stankevicius E. Local Vibrational Therapy for Essential Tremor Reduction: A Clinical Study. Medicina (Kaunas). 2020 Oct 21;56(10):552. doi: 10.3390/medicina56100552. PMID 33096872